CLINICAL TRIAL: NCT04624269
Title: A Multicenter, Double-blind, Randomized and Parallel Controlled Study of Hydroxychloroquine Sulfate in the Treatment of Recurrent Miscarriage With Antiphospholipid Syndrome
Brief Title: A Study of Hydroxychloroquine Sulfate in the Treatment of Recurrent Spontaneous Abortion With Antiphospholipid Syndrome
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai First Maternity and Infant Hospital (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other); Fudan University (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Provincial Tongde Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShanghaiFMIH-HCQ
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Antiphospholipid Syndrome; Recurrent Miscarriage
Keywords: Antiphospholipid syndrome; hydroxychloroquine; Recurrent Miscarriage
MeSH Terms: conditions — Antiphospholipid Syndrome; Abortion, Habitual | interventions — Hydroxychloroquine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hydroxychloroquine sulfate Tablets (Experimental): drug:Hydroxychloroquine sulfate Tablets,0.1mg bid po
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets
- placebo (Placebo Comparator): drug:placebo,0.1mg bid po
  Interventions: Drug: Hydroxychloroquine Sulfate Tablets

INTERVENTIONS:
Drug: Hydroxychloroquine Sulfate Tablets — Hydroxychloroquine Sulfate Tablets ,0.1mg，bid po
  Other Names: Fenle

SUMMARY:
The efficacy of low-dose aspirin combined with low-molecular-weight heparin treatment for improving antiphospholipid syndrome and maternal-fetal outcome of patients is recognized by various countries and recommended by the guidelines. However, there are still 20-30% of APS patients whose treatment fails. Therefore, the standard treatment effect is still not ideal, and other treatment options need to be explored. The purpose of this study is to conduct a randomized double-blind, parallel controlled study of patients with recurrent miscarriage and APS in addition to standard treatment, plus hydroxychloroquine sulfate (HCQ) or placebo, to observe the effects of HCQ on pregnancy outcome in patients with abortion and APS, to evaluate the effectiveness and safety of HCQ treatment.

DETAILED DESCRIPTION:
This study uses a multi-center, double-blind, randomized, parallel-controlled research model. In addition to the standard anticoagulant drugs for antiphospholipid syndrome, patients with recurrent miscarriage and APS who meet the enrollment criteria will be randomly divided into hydroxychloroquine sulfate( HCQ) group or placebo group, and randomly assigned according to a 1:1 ratio. Observe the efficacy and safety.

The Hydroxychloroquine sulfate(HCQ) group is the test group. Hydroxychloroquine sulfate 0.2g/d (sig: 0.1g bid po) will be applied 3 months before pregnancy, pregnancy will be started at the 4th month, and aspirin 50mg/d will be added after menstruation( sig: 25mg bid po), low molecular weight heparin 4000-6000 U/d after ovulation or 1 week before embryo transplantation; the placebo group is the control group, and placebo 0.2g/d (sig: 0.1 g bid po) from the fourth month of pregnancy, add aspirin 50mg/d (sig: 25mg bid po) after menstruation, and add low molecular heparin 4000-6000 U/d after ovulation or 1 week before embryo transplantation Both groups were followed up by telephone every 1 month to obtain medication compliance, whether there were adverse reactions, etc., and both oth groups were followed up every 3 months for non-pregnant women by outpatient service , until pregnancy. If the patient is not pregnant within one year, The clinical study of this patient will be terminated, and the patients will be followed up for adverse reactions by telephone one month and three months after withdrawal. If you are pregnant, follow up in the first trimester immediately, and arrange a follow-up every three months thereafter (defined as follow-up in the first trimester, follow-up in the second trimester and follow-up in the third trimester). The drug was discontinued on the day of delivery and the postpartum follow-up was completed 6 weeks after delivery. So, therefore, the entire study time is approximately 27 months.

The researcher mainly records the subjects' vital signs, laboratory indicators, adverse events and combined medications, as well as related indicators of pregnancy check-ups (such as uterine artery blood flow, presence or absence of pregnancy complications, fetal complications, etc.)

ELIGIBILITY:
Inclusion Criteria:

* Patients who want to conceive，with recurrent miscarriage and antiphospholipid syndrome (APS) .
* Agree to join the study and sign the informed consent of the study.

Exclusion Criteria:

* Women who are already pregnant.
* Allergies or adverse events to Hydroxychloroquine(HCQ),such as allergies to the active substance -aminoquinoline or allergies to HCQ or any other chemical components of placebo.
* Patients with any changes in the retina or visual field caused by treatment with 4-aminoquinoline compounds;
* HCQ is currently being used
* Weight <45kg
* Psoriasis
* Uncontrolled epilepsy
* Anti-ENA antibody positive
* Renal replacement therapy
* Other serious active complications (human immunodeficiency virus, hepatitis B)
* Porphyria
* History of retinopathy
* History of galactose intolerance, history of lactase deficiency, or history of glucose-galactose malabsorption
* Participate in any other clinical trial drug research at the same time.
* Previous treatment failure with Hydroxychloroquin
* Others: such as poor compliance, or those who cannot be followed up on schedule due to certain factors.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 384 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Hydroxychloroquine can improve the pregnancy outcome of patients with recurrent miscarriage and antiphospholipid syndrome | 16 weeks
  Hydroxychloroquine is associated with successful pregnancy outcome at 12 weeks of gestation

SECONDARY OUTCOMES:
Hydroxychloroquine can reduce the occurrence of complications during pregnancy | 27 weeks
  Reduced incidence of major adverse pregnancy outcomes related to antiphospholipid syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Bao shihua, doctor, Study Chair — shanghai First Maternity and Infant Hospital, Tongji University School of Medicin
Locations (1):
- shanghai First Maternity and Infant Hospital, Tongji University School of Medicin, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak A, Cheung MW, Cheak AA, Ho RC. Combination of heparin and aspirin is superior to aspirin alone in enhancing live births in patients with recurrent pregnancy loss and positive anti-phospholipid antibodies: a meta-analysis of randomized controlled trials and meta-regression. Rheumatology (Oxford). 2010 Feb;49(2):281-8. doi: 10.1093/rheumatology/kep373. Epub 2009 Dec 4. PMID 19965971
- [Result] Sciascia S, Branch DW, Levy RA, Middeldorp S, Pavord S, Roccatello D, Ruiz-Irastorza G, Tincani A, Khamashta M, Schreiber K, Hunt BJ. The efficacy of hydroxychloroquine in altering pregnancy outcome in women with antiphospholipid antibodies. Evidence and clinical judgment. Thromb Haemost. 2016 Jan;115(2):285-90. doi: 10.1160/TH15-06-0491. Epub 2015 Sep 17. PMID 26421409
- [Result] Abarientos C, Sperber K, Shapiro DL, Aronow WS, Chao CP, Ash JY. Hydroxychloroquine in systemic lupus erythematosus and rheumatoid arthritis and its safety in pregnancy. Expert Opin Drug Saf. 2011 Sep;10(5):705-14. doi: 10.1517/14740338.2011.566555. Epub 2011 Mar 22. PMID 21417950
- [Result] Mekinian A, Lazzaroni MG, Kuzenko A, Alijotas-Reig J, Ruffatti A, Levy P, Canti V, Bremme K, Bezanahary H, Bertero T, Dhote R, Maurier F, Andreoli L, Benbara A, Tigazin A, Carbillon L, Nicaise-Roland P, Tincani A, Fain O; SNFMI and the European Forum on Antiphospholipid Antibodies. The efficacy of hydroxychloroquine for obstetrical outcome in anti-phospholipid syndrome: Data from a European multicenter retrospective study. Autoimmun Rev. 2015 Jun;14(6):498-502. doi: 10.1016/j.autrev.2015.01.012. Epub 2015 Jan 21. PMID 25617818
- [Result] Branch DW, Peaceman AM, Druzin M, Silver RK, El-Sayed Y, Silver RM, Esplin MS, Spinnato J, Harger J. A multicenter, placebo-controlled pilot study of intravenous immune globulin treatment of antiphospholipid syndrome during pregnancy. The Pregnancy Loss Study Group. Am J Obstet Gynecol. 2000 Jan;182(1 Pt 1):122-7. doi: 10.1016/s0002-9378(00)70500-x. PMID 10649166
- [Result] Sciascia S, Hunt BJ, Talavera-Garcia E, Lliso G, Khamashta MA, Cuadrado MJ. The impact of hydroxychloroquine treatment on pregnancy outcome in women with antiphospholipid antibodies. Am J Obstet Gynecol. 2016 Feb;214(2):273.e1-273.e8. doi: 10.1016/j.ajog.2015.09.078. Epub 2015 Sep 30. PMID 26429521